CLINICAL TRIAL: NCT05339945
Title: Towards an Early Integration of Palliative Care in Oncology: Descriptive Study of Needs for Patients With Metastatic Cancer and the Adequacy of These Needs With Healthcare Facilities
Brief Title: Towards an Early Integration of Palliative Care in Oncology
Acronym: BESACE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210724; 2021-A01007-34 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-04-06; First posted 2022-04-21 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Cancer; Palliatives Treatments
Keywords: metastatic cancer; palliative care; oncology; health needs; early integration
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the study is to describe the nature and to estimate the prevalence the health needs of patients with metastatic cancer and their main caregivers, between the period from diagnosis to death.

As secondary objectives, the study aims:

* to determinate the proportion of patients with an indication for palliative care according to Hui et al., and to describe the adequation of health needs and the services for them;
* to study the association between clinical pathway and the indication of targeted palliative care;
* to study the association between the integration of palliative care service and the adequation of health needs service of patients;
* to study the factors such as the disease, the practice and the care, contribute to the patient's survivor of 1 year.

DETAILED DESCRIPTION:
This is a descriptive, transversal, multicenter study, which will be performed in healthcare facilities in Ile de France area.

Each investigator center will be composed by oncologist / palliative care and support team. 10 centers will participate to the study, enrollement will be perfomed during 6 months targetting 400 patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years;
* Diagnosed metastatic cancer;
* Outpatient or inpatient care at a participating site to the study;
* Affiliation to the social security scheme;
* Patient informed and non-opposed to participate to the study.

Exclusion Criteria:

* Testicular or choriocarcinoma ovarian cancer;
* Hematology cancer;
* No understanding french language;
* Unable to express if needed his non-opposition opinion, according to physician investigator;
* Visually impaired, hearing impaired or aphasic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with diagnosed metastatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Auto-evaluation | at baseline
  Evaluation by patient and principal caregiver the health needs.
  Questionnaires: EORTC-QLQ C30
Auto-evaluation | at baseline
  Evaluation by patient and principal caregiver the health needs.
  Questionnaires: SCNS-SF34
Auto-evaluation | at baseline
  Evaluation by patient and principal caregiver the health needs.
  Questionnaires: EPICES
Auto-evaluation | at baseline
  Evaluation by patient and principal caregiver the health needs.
  Questionnaires: Echelle de Zarit.

SECONDARY OUTCOMES:
Description of disease | at baseline
Clinical trajectory description | at baseline
Proportion (%) of patients needing palliative treatment | at the end of study
Survivor (%) | at 1 year
  Vital statute of patients at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marine SAHUT D'IZARN, MD, Principal Investigator — Mobile palliative care and support team, Ambroise Paré hospital, APHP
Locations (1):
- Mobile palliative care and support team, Ambroise Paré hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hui D, Mori M, Watanabe SM, Caraceni A, Strasser F, Saarto T, Cherny N, Glare P, Kaasa S, Bruera E. Referral criteria for outpatient specialty palliative cancer care: an international consensus. Lancet Oncol. 2016 Dec;17(12):e552-e559. doi: 10.1016/S1470-2045(16)30577-0. PMID 27924753
- [Derived] Sahut d'Izarn M, Vinant P, Bouleuc C, Joffin I, Vincent B, Barth C, Serresse L, Codogno A, Behal F, Ya-de Rauglaudre L, Jacota M, Gassama M, de Stampa M. Healthcare needs of patients with metastatic cancer and impacts of social vulnerability: a multicentric cross-sectional study in France. BMC Palliat Care. 2025 Sep 29;24(1):233. doi: 10.1186/s12904-025-01882-4. PMID 41024046